CLINICAL TRIAL: NCT07196345
Title: Efficacy and Safety of Trifluridine/Tipiracil Combined With Radiotherapy in Elderly Patients With Locally Advanced Esophageal Cancer
Brief Title: TAS-102 Plus Radiotherapy in Elderly ESCC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jiandong Zhang, Director of Department of Radiotherapy, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2025(055)
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ESCC; TAS 102; Radiotherapy
MeSH Terms: interventions — trifluridine tipiracil drug combination; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-102 + Radiotherapy (Experimental)
  Interventions: Drug: TAS-102; Radiation: Radiotherapy

INTERVENTIONS:
Drug: TAS-102 — Administered orally at 35 mg/m²/dose twice daily (morning and evening), in a bi-weekly regimen on Days 1-5.
Radiation: Radiotherapy — Total dose of 50-60 Gy, delivered in 25-28 fractions, administered Monday through Friday (daily) until the full prescribed dose is achieved.

SUMMARY:
This study is a single-arm, multicenter clinical trial evaluating the efficacy and safety of radiotherapy combined with TAS-102 monotherapy in elderly patients with locally advanced esophageal cancer.

Treatment Phase: The treatment phase is divided into a Phase I stage and a Phase II stage. The Phase I stage aims to explore the maximum tolerated dose (MTD) of TAS-102 in elderly esophageal cancer patients. A total of 9 subjects were enrolled, and the dose was escalated from 30 mg/m² in 5 mg/m² increments up to 40 mg/m². The MTD was defined as the highest drug dose at which no dose-limiting toxicity (DLT) was observed in more than 40% of treated patients during the first two weeks of combined radiotherapy and TAS-102 administration. The Phase II stage aims to investigate the efficacy of radiotherapy combined with TAS-102 at the MTD in elderly esophageal cancer patients, with 36 subjects enrolled.

Consolidation Phase: Following the treatment phase, subjects had a 3-4 week rest period. This was followed by consolidation therapy with TAS-102 monotherapy at a dose of 35 mg/m², administered twice daily on days 1-5 of a 28-day cycle for two cycles.

Subsequently, patients entered the efficacy and safety follow-up phase until the study endpoints were reached or after a full 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly confirmed histologically or cytologically diagnosed esophageal squamous cell carcinoma.
* Age between 65 and 85 years.
* Esophageal cancer staged as IIB to IVB according to the 8th edition AJCC staging system (including IVB with supraclavicular or celiac lymph node metastasis, but excluding IVB with other distant metastases).
* ECOG performance status of 0 or 1.
* No history of esophageal perforation, active esophageal bleeding, or significant invasion of the trachea or major thoracic blood vessels.
* No prior anticancer therapy such as radiotherapy or chemotherapy. Adequate bone marrow function: hemoglobin ≥9 g/dL, white blood cells ≥3.0×10⁹/L, neutrophils ≥1.5×10⁹/L, platelets ≥100×10⁹/L.
* Adequate liver and kidney function: serum creatinine (Scr) ≤1.5×ULN, total bilirubin ≤1.5×ULN, ALT and AST ≤2.5×ULN.
* No history of interstitial lung disease.
* Forced expiratory volume (FEV1) ≥0.8 liters.
* Signed informed consent form before study initiation.

Exclusion Criteria:

* Patients with hematogenous metastasis or distant lymph node metastasis (except supraclavicular or celiac lymph node metastasis), multiple esophageal cancer lesions, or malignant pleural/pericardial effusion.
* History of radiotherapy, chemotherapy, or surgery targeting the primary tumor or lymph nodes.
* Tracheoesophageal fistula, invasion of the trachea or main bronchi by the primary tumor, deep esophageal ulcer, or hematemesis.
* Severe comorbidities such as active infection, cardiovascular disease, or pulmonary disease.
* History of other malignancies except adequately treated non-melanoma skin cancer.
* Participation in another clinical trial within the past 30 days.
* Any other condition deemed by the investigator to preclude participation in the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-09-25 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-years OS rate | Approximately 24 months after the last subject participating in
  The percentage of study participants who are still alive at 2 years after the starting date of the study drug, calculated from the starting date of the study drug to the date of death from any cause.

SECONDARY OUTCOMES:
ORR | Approximately 4 months after the last subject participating in
  The time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
PFS | Approximately 12 months after the last subject participating in
  The time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first (per RECIST 1.1).
Adverse Event (AE) | Up to approximately 2 years
  Type, incidence, grading (based on NCI-CTCAE v5.0 criteria), and duration of adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China